CLINICAL TRIAL: NCT02014493
Title: Respiratory Effort in Preterm Infants in the Transition From Continuous Positive Airway Pressure (CPAP) to High Flow Nasal Cannulae (HFNC)
Brief Title: Changes in Respiratory Effort in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HHB-2013
Record Dates: First submitted 2013-12-04; First posted 2013-12-18 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Premature Birth
Keywords: Respiration; Noninvasive Ventilation; Work of breathing; Infant, premature; Electromyography; Diaphragm
MeSH Terms: conditions — Premature Birth; Respiratory Aspiration | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFNC first (Active Comparator): 4 hours with High Flow Nasal Cannulae (HFNC) 6 l/pr.min, then 4 hours with Continuous Positive Airway Pressure (CPAP) 6l/pr.min.
  Interventions: Procedure: High Flow Nasal Cannulae (HFNC)
- CPAP first (Active Comparator): 4 hours Continuous Positive Airway Pressure (CPAP) 6 l/pr.min, then 4 hours High Flow Nasal Cannulae (HFNC) 6 l/pr.min.
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: High Flow Nasal Cannulae (HFNC) — HFNC 6 l/pr.min
  Arms: HFNC first
Procedure: Continuous Positive Airway Pressure (CPAP) — CPAP 6 l/pr.min
  Arms: CPAP first

SUMMARY:
Continuous Positive Airway Pressure (CPAP) is used to treat preterm infants with an immature respiratory center and having respiratory distress. CPAP requires intensive care monitoring and special qualified staff. Continuous positive pressure makes a constant noise around the child and can lead to an uncomfortable environment.The fixture of the binasal prongs can cause nasal trauma after to tight attachment.Minimizing the time on CPAP is considered important for the child.

Recently High-Flow Nasal Cannula (HFNC) has become widely used in modern newborn intensive care units.HFNC is considered to be easy to apply and a more comfortable respiratory support for the preterm infant with mild and moderate respiratory distress. HFNC gives warm humified air with high flow through a nasal cannulae. HFNC is used as part of withdrawal from intensive respiratory support, to prevent respiratory distress and as a respiratory support after extubation.

There is still uncertainty about safety and effectiveness of HFNC. The aim of this study is to investigate the preterm infants respiratory effort by measuring electrical activity in diaphragm (Edi max and Edi min), respiratory parameters and a clinical observation using a scoring system inspired by Silverman- Andersen retraction score. It is expected that measured electrical activity in the diaphragm, measured respiratory parameters combined with bedside observations provide applicable knowledge about preterm infants respiratory effort in transition from CPAP to HFNC.

DETAILED DESCRIPTION:
Data material will be stored on a separate computer in a sheltered home Directory. All data will be anonymous. Edi signals are transported from Servo-I ventilator with neural access through a communication port to a personal computer.Respiratory parameters will be stored in Picis (High Performance Hospital Information System). For the Statistical analyzes a T-test will be carried out, and data from the pilot study will decide the power to see whether we reject or retain the 0 hypothesis: " There are no changes in the preterm infants respiratory effort in transition from CPAP to HFNC".

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who are stable on Nasal Continuous Positive Airway Pressure (nCPAP) with flow 8l/min
* <34 and >28 gestational weeks, respiratory stable last 72 hours.
* 1 kilo
* Fi02< 30%
* C02<9
* written informed consent by parents/caregivers

Exclusion Criteria:

* need for sedation
* damage on the phrenic nerve
* anomalies in the upper airways

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neural control of respiration | 4 months
  reflected by electrical activity of the diaphragm (Edi): inspiratory drive (Edi peak) and tonic activity (Edi min). A nasogastric feeding tube with ten microsensors will measure action potentials from the phrenic nerve to the diaphragm.

SECONDARY OUTCOMES:
Respiratory signs | 4 months
  Observation scale inspired by Silverman- Anderson retraction score. Observation of chest movement, intercostal retraction and xiphoid retraction.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Bergseng, MD PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- Newborn Intensive Care Unit, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Brenne H, Grunewaldt KH, Follestad T, Bergseng H. A randomised cross-over study showed no difference in diaphragm activity during weaning from respiratory support. Acta Paediatr. 2018 Oct;107(10):1726-1732. doi: 10.1111/apa.14303. Epub 2018 Apr 4. PMID 29504671